CLINICAL TRIAL: NCT01535339
Title: Evaluating a Novel Method of EEG Evoked Response Potential Analysis in Sport Concussion Assessment - Test Stability and Effect of Concussion
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-03
Record Dates: First submitted 2012-02-12; First posted 2012-02-17 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mild Traumatic Brain Injury; mTBI; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Phase I - Normative: Athletes who does not participate in contact sport with no recent concussion
- Phase IIa - Concussed: Athletes with recent concussion
- Phase IIa - Control: Athletes with no recent concussion
- Phase IIb - Athletes: Athletes with no recent concussion

SUMMARY:
Mild traumatic brain injury (mTBI), also known as concussion, occurs commonly in sport. Despite ongoing research, there is no highly sensitive clinical test for cognitive function. This makes the clinical diagnosis of concussion particularly difficult as the clinical presentation of concussion is highly variable with symptoms often evolving over time. Given the variability in concussion presentations, there is no single test that can diagnose a concussion. Current recommendations are that sports medicine providers apply a multifaceted concussion assessment battery that combines subjective symptoms, motor control and cognitive assessment.

This investigation is designed to evaluate the clinical utility of ElMindA's BNA scores in detecting and managing concussive injuries. This study will establish the reliability of BNA™ scores over clinically relevant assessment intervals and investigate the effect of SRC and sub-concussive head impacts on BNA scores.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Aged 14-26 years
* Enrolled in a recognized high school or college
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self)
* Currently participate in a non-contact sport.
* Member of an organized athletic team or regularly train for and participate in independent athletic contests during at least one sports season.
* Right handed subject

Exclusion Criteria:

* Currently participate in a contact sport.
* Bald or has dread locks/long and thick hair.
* Any diagnosed psychiatric disorder
* History of CNS injury or disease
* Any neuropsychological disorders
* History of learning disability.
* History of any medication affecting CNS.
* Active head lice infection, open scalp wound, deafness or/and blindness.
* Sustained a diagnosed concussion within the previous 6 months

Phase 2a:

Inclusion Criteria:

* Aged 14-26 years.
* For Arm 1: Within 1 week post-concussion (sports-related).
* For Arm 1: Currently symptomatic
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self).
* Member of an organized athletic team or regularly train.
* Enrolled in a high school or college.

Exclusion Criteria:

* Bald or has dread locks/long and thick hair.
* Current or history of ADHD.
* Active head lice infection, open scalp wound, deafness or/and blindness.
* Sustained a concussion within the past 6 months.
* Current or history of moderate or severe TBI, any brain injury with positive neuroimaging findings, or brain surgery.

Phase 2b:

Inclusion Criteria:

* Aged 14-26 years.
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self).
* Member of a contact sport team which carries out head impact monitoring over the course of the playing season.
* Enrolled in a high school or college.

Exclusion Criteria:

* Bald or has dread locks/long and thick hair.
* Current or history of ADHD.
* Active head lice infection, open scalp wound, deafness or/and blindness.
* Sustained a concussion within the past 6 months.
* Current or history of moderate or severe TBI, any brain injury with positive neuroimaging findings, or brain surgery.
* Any diagnosed psychiatric disorder.
* History of CNS injury or disease
* Any neuropsychological disorders.
* History of learning disability.
* History of any medication affecting CNS.

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Phase 1: gender-balanced groups of 30 healthy high school (14-17 years old) and 30 healthy college aged (18-26 years old) individuals who participate in non-contact sports Phase 2a: 30 high school and/or collegiate athletes aged 14-26 years with concussion and 30 matched control athletes.
  Phase 2b: at least 30 high school and/or collegiate contact sport athletes aged 14-26 years whose head impacts are monitored during games and practices.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of Brain Network Activation(BNA™)Scores | P.I - days 0 , 7, 42, 365 ; P.IIa - 1 week of injury, 48 hours of symptom resolution, 48 hours of clearance to sport, 1 month after symptom resolution; P.IIb - baseline, mid season, 30 days of completion of the season

SECONDARY OUTCOMES:
Correlation Of The Change In BNA™ Scores To Clinical Diagnstic | P.I - days 0 , 7, 42, 365 ; P.IIa - 1 week of injury, 48 hours of symptom resolution, 48 hours of clearance to sport, 1 month after symptom resolution; P.IIb - baseline, mid season, 30 days of completion of the season
Correlation Of The Change In BNA™ Scores To Neurocognitive Tests Scroes | P.IIa - 1 week of injury, 48 hours of symptom resolution, 48 hours of clearance to sport, 1 month after symptom resolution; P.IIb - baseline, mid season, 30 days of completion of the season
Correlation Of The Change In BNA™ Scores To Reaction Time Scores | P.IIa - 1 week of injury, 48 hours of symptom resolution, 48 hours of clearance to sport, 1 month after symptom resolution; P.IIb - baseline, mid season, 30 days of completion of the season

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan NeuroSport Concussion Program, Ann Arbor, Michigan, United States